CLINICAL TRIAL: NCT02088658
Title: Technology Intensified Diabetes Education Study in African Americans With Type 2 Diabetes
Brief Title: Technology Intensified Diabetes Education Study in African Americans
Acronym: TIDES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Medical University of South Carolina (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00015064; 1R01DK098529 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Type II; African Americans; Blacks; non-Hispanic Blacks; Randomized Control Trial; Controlled Clinical Trial; Behavioral Research; Behavioral Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Techonology Intensified (Experimental): Subjects randomized to this group will receive: 1) the FORA system for self-monitoring; 2) weekly telephone-delivered diabetes education/skills training; 3) patient activation (list of 5 questions to ask their provider at every visit and training on how to ask the questions); and 4) patient empowerment (diabetes responsibility contracts, personal goals, and flow charts for patients to record lab results/medications and training on how to use the empowerment tools). The intervention will be delivered by telephone once a week for 12 weeks with each session lasting ~30 minutes.
  Interventions: Behavioral: Technology Intensified
- Usual Care (No Intervention): Apart from study visits, patients will be followed by their primary care providers. The provider will be responsible for determining treatment parameters, making changes in the treatment regimen, and determining the timing of follow up visits. Between scheduled office encounters, contact between patient and provider will be patient initiated. The provider may use clinic nurses to follow up on problematic patients or patients with abnormal results. In essence, this group will receive the current standard of care at the study clinics.

INTERVENTIONS:
Behavioral: Technology Intensified — The intervention is based on the Information-Motivation-Behavioral Skills (IMB) model and provides information, motivation, and behavioral skills training (using motivational enhancement techniques). Patients will be assigned the FORA 2-in-1 Telehealth System and provided glucose test strips to allow testing at least once a day. They will be asked to perform glucose testing and blood pressure measurement using the FORA system once daily. They will be asked to upload the measurements daily as soon as possible after the test is performed. The nurse educators will have access to a secure server to which the uploaded measurements are stored in real time. The glucose and BP readings will be used to tailor and reinforce behavior change during weekly telephone-delivered diabetes education sessions.
  Arms: Techonology Intensified

SUMMARY:
The purpose of this study is to test the usefulness of an intervention that combines technology with diabetes education and skills training. This study has been designed specifically for African Americans with poorly controlled type 2 diabetes.

DETAILED DESCRIPTION:
African Americans (AA) with type 2 diabetes (T2DM) have higher prevalence of diabetes, poorer metabolic control (i.e. poorer blood glucose, blood pressure, and lipid control), and greater risk for complications and death compared to White Americans. Hemoglobin A1c (HbA1c) is the primary marker for glycemic control and is a strong independent predictor of development of complications and increased mortality in T2DM. Key self-care behaviors that influence glycemic control (and HbA1c) include diet, physical activity, self-monitoring of blood glucose and medication adherence. Systematic review of multiple randomized clinical trials (RCTs) show that self-care interventions that include diabetes education and skills training are effective in improving metabolic control in diabetes. Recent findings indicate that patients with diabetes, especially ethnic minority patients, prefer telephone-delivered diabetes education to group visits or internet-based education. Multiple RCTs have documented the effectiveness of telephone-delivered self-care interventions in T2DM. Preliminary data from our group also suggest that a culturally-tailored telephone-delivered diabetes education and skills training intervention is an effective strategy to improve metabolic control in AA patients with T2DM.

This study provides a unique opportunity to address gaps in the literature by testing the efficacy of a technology-intensified diabetes education/skills training (TIDES) intervention in AAs with poorly controlled T2DM. The long-term goal of the project is to identify effective strategies to improve metabolic control and hence reduce diabetes complications and mortality rates in AAs with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Clinical diagnosis of T2DM and HbA1c ≥8% at the screening visit
* Self-identified as AA
* Subject must be willing to use the FORA monitoring system for 12 months
* Subjects must be able to communicate in English
* Subjects must have access to a telephone (landline for data uploads) for the study period

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Participation in other diabetes clinical trials
* Alcohol or drug abuse/dependency
* Active psychosis or acute mental disorder
* Life expectancy <12 months

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 months post randomization
  Hemoglobin A1c (HbA1c): blood specimens will be collected at the screening visit, as well as the 3-months, 6-months, 9-months, and 12-months follow-up visits

SECONDARY OUTCOMES:
Blood Pressure | 12 months post randomization
  Blood pressure measurement: Blood pressure readings will be obtained at baseline, 3-months, 6-months, 9-months, and 12-months, following the American Heart Association guidelines. The device will be programmed to take 3 readings at 2 minute intervals, and give an average of the 3 blood pressure readings.
Resource Utilization & Cost | 12 months post randomization
  Resource Utilization & Cost: Information on hospitalizations, physician/professional visits, and medications will be captured.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Williams JS, Lynch CP, Knapp RG, Egede LE. Technology-Intensified Diabetes Education Study (TIDES) in African Americans with type 2 diabetes: study protocol for a randomized controlled trial. Trials. 2014 Nov 25;15:460. doi: 10.1186/1745-6215-15-460. PMID 25425504

DOCUMENTS (1):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02088658/Prot_001.pdf